CLINICAL TRIAL: NCT04100785
Title: A Pilot Investigation of Clinician-guided Internet-Delivered Cognitive Behavioural Therapy for Depressed Patients in an Outpatient Hospital Setting
Brief Title: A Pilot Investigation of Clinician-guided Internet-Delivered Cognitive Behavioural Therapy for Depressed Patients
Acronym: iCBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mental Health, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015/00404
Record Dates: First submitted 2019-09-16; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-delivered Cognitive Behavioural Therapy (iCBT) (Experimental): The iCBT programme comprised of 6 online modules, delivered over 4 weeks, with 3 face-to-face sessions provided by a clinician.The face-to-face sessions were conducted at week 1, 3 and 4. The objectives of the face-to-face sessions was for participants to discuss with the clinician about the application of the content of the modules and the active therapeutic interventions were all found in the online modules.
  Interventions: Behavioral: Internet-delivered Cognitive Behavioural Therapy
- Delayed Wait-list control (No Intervention): The delayed wait-list control did not receive any therapy interventions for 4 weeks from the pre-treatment assessment and from the fifth week onwards, they received the same intervention as the iCBT experimental group.

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive Behavioural Therapy — The iCBT programme comprised on 6 online modules. Module 1 provided an introduction to the symptoms of depression, its causes and information on CBT. Module 2 covered problem-solving strategies. Module 3 provided information on problematic thought patterns and beliefs in depression. Module 4 entailed identifying problematic thought patterns and using various techniques to counter problematic thoughts. Module 5 covered pleasurable activities scheduling to help increase activity levels.
  Arms: Internet-delivered Cognitive Behavioural Therapy (iCBT)

SUMMARY:
This study aims to explore the efficacy and acceptability of a clinician-guided internet-based Cognitive Behavioural Therapy (iCBT) programme for patients with depression, in Singapore.

DETAILED DESCRIPTION:
All outpatients, from the Institute of Mental Health, Singapore, who are diagnosed with a primary diagosis of mild to moderate depression and were referred to the Psychology Department for therapy were invited to take part in this research. Participants were randomised into two groups: iCBT Intervention Group and Delayed Waitlist-Control Group. The four-week iCBT programme comprised of three face to face 30-minute sessions with a clinician and six online modules).The treatment group is hypothesised to exhibit pre-post improvements in depressive symptoms, compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 65 years old
* Not currently seeing a therapist for any form of invidual or group therapy
* Diagnosed with a primary diagnosis of depression by IMH psychiatrist
* A total score of above 9 on the Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001), indicating at least mild symptoms
* If using medication for depression then on a stable dose for at least 1 month,
* Provides informed consent
* Able to read and speak at least Primary 6 level English
* Adequate IT skills to operate iCBT programme

Exclusion Criteria:

* Severe depression (i.e. score = 23 on PHQ-9)
* Strong suicidal ideation (i.e. score > 2 on Question 9 of the PHQ-9)
* Current active suicidal intention or plan
* Presenting problem is not depression
* Does not meet the minimum English language requirements stated above
* Participants who are concurrently attending other forms of group/individual psychotherapy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-08-09 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-16 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ9) | week 1, week 3, week 4 and 3-month follow-up
  The PHQ-9 is a nine-item self-report measure of symptoms and severity of major depressive disorder, based on the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV; American Psychiatric Association, 2000) criteria for Major Depressive Disorder. Scores on each item range from 0 (not at all) to 3 (nearly every day). An overall cut-off score of 10 or greater has been found to be sensitive to a DSM-IV diagnosis of depression (Kroenke, Spitzer, Williams, amp; Löwe, 2010). The PHQ9 has an internal reliability of 0.86- 0.89, sensitivity of 88% and specificity of 88% for the clinical cut-off of 10. Test-retest reliability of 0.84, and moderately correlated(r=0.58) with the SF-20 mental health scale. (Kronke et al.,2001).

SECONDARY OUTCOMES:
Change in Generalised Anxiety Disorder-7 (GAD-7) | week 1, week 3, week 4 and 3-month follow-up
  The GAD-7 is a seven-item self-report measure of symptoms and severity of Generalised Anxiety Disorder (GAD), based on the DSM-IV criteria for GAD. Scores for each item range from 0 (not at all) to 3 (nearly every day). An overall cut-off score of 10 or greater has been found to be sensitive to DSM-IV diagnoses of GAD, social phobia and panic disorders (Kroenke, Spitzer, Williams, Monahan, amp; Lo ̈we, 2007). The GAD-7 has an internal reliability of 0.92, test-retest reliability of 0.83, and criterion validity of 0.75 with SF-20 mental health scale (Spitzer et al., 2006) .The GAD-7 is increasingly adopted in empirical studies and in large scale dissemination studies as a general measure of shifts in anxiety symptoms (Clark et al., 2009).
Change in Work and Social Adjustment Scale (WSAS) | week 1, week 3, week 4 and 3-month follow-up
  The WSAS is a five-item self-report measure of the extent of impairment in work and social functioning. Scores ranged from 0 to 40. An overall score of above 20 appears to suggest moderately severe or worse psychopathology. Scores between 10 and 20 are associated with significant functional impairment but less severe clinical symptomatology. The WSAS has an internal reliability of 0.70-0.94, Test-retest reliability of 0.73. Convergent validity compared with clinical interviews and severity of depression is 0.76-0.86.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon HX Lu, DPsych, Principal Investigator — Institute of Mental Health, Singapore